CLINICAL TRIAL: NCT01563952
Title: Impact of IVUS-guided Chronic Total Occlusion InterVention With DrUg-eluting Stents on Mid-term Angiographic and Clinical Outcomes (CTO-IVUS Study)
Brief Title: Impact of Intravascular Ultrasound(IVUS)-Guided Chronic Total Occlusion Intervention With Drug-eluting Stents
Acronym: CTO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yangsoo Jang, Professor of cardiology, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2010-0023
Record Dates: First submitted 2012-03-12; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non-IVUS guided endeavor-R group (Active Comparator): 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Interventions: Device: Non-IVUS guided intervention with Endeavor Resolute stent (zotarolimus-eluting stent, Medtronic)
- IVUS guided endeavor-R group (Experimental): 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Interventions: Device: IVUS guided intervention with Endeavor Resolute stent (zotarolimus-eluting stent, Medtronic)
- Non-IVUS guided Nobori group (Active Comparator): 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Interventions: Device: Non-IVUS guided intervention with Nobori stent (biolimus A9-eluting stent, Terumo)
- IVUS guided Nobori group (Experimental): 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Interventions: Device: IVUS guided intervention with Nobori stent (biolimus A9-eluting stent, Terumo)

INTERVENTIONS:
Device: Non-IVUS guided intervention with Endeavor Resolute stent (zotarolimus-eluting stent, Medtronic) — 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Arms: Non-IVUS guided endeavor-R group
Device: IVUS guided intervention with Endeavor Resolute stent (zotarolimus-eluting stent, Medtronic) — 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Arms: IVUS guided endeavor-R group
Device: Non-IVUS guided intervention with Nobori stent (biolimus A9-eluting stent, Terumo) — 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Arms: Non-IVUS guided Nobori group
Device: IVUS guided intervention with Nobori stent (biolimus A9-eluting stent, Terumo) — 2x2 randomization by the treatment of IVUS-guided intervention vs. Non-IVUS guided intervention and the types of the implanted DES, Endeavor-R vs. Nobori.
  Arms: IVUS guided Nobori group

SUMMARY:
Guidance of stenting by IVUS has been proposed as a method to reduce restenosis rates, because lumen and stent dimensions can be accurately determined by intravascular ultrasound (IVUS).

DETAILED DESCRIPTION:
Guidance of stenting by IVUS has been proposed as a method to reduce restenosis rates, because lumen and stent dimensions can be accurately determined by intravascular ultrasound (IVUS). However, randomized studies investigating this strategy have yielded inconsistent results. Therefore, the investigators hypothesized that the potential advantages of IVUS guidance would be most apparent in Chronic Total Occlusion (CTO) intervention and try to evaluate the impact of IVUS-guided chronic total occlusion intervention with drug-eluting stents on mid-term angiographic, IVUS and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 20 years or ≤ 80 years old
2. On coronary angiography, complete obstruction of coronary blood flow (TIMI grade 0) with estimated occlusion duration ≥ 3months.
3. On coronary angiography, Reference vessel diameter of 2.5 to 4.0mm by operator assessment
4. On coronary angiography, Total length of total occluded lesion and main lesion is less than 80mm and lesions can be treated less than 4 stents.
5. Guide wire can be passed through occluded lesion without complications
6. Patients who can keep the dual antiplatelet treatment (aspirin, clopidogrel) more than 6 months after procedure

Exclusion Criteria:

1. Hypersensitivity reaction or side effects to Aspirin, Clopidogrel, Biolimus A9 and Zotarolimus
2. unprotected Left main disease
3. Cardiogenic shock or LV ejection fraction ≤ 30%
4. Previous stent restenotic lesion
5. Treated within 2 weeks at the same lesion.
6. Creatinine level ≥ 2.0 mg/dL or ESRD
7. Severe tortuous and calcified lesion (Unobtainable IVUS image)
8. Life expectancy < 1 year
9. Severe hepatic dysfunction (3 times normal reference values)
10. Pregnant women or women with potential childbearing

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
event rate of cardiac death within 12 months | 12 months after CTO intervention.
  Between IVUS guided intervention and non-IVUS guided intervention in patient with chronic total occlusion, the difference of post-procedural success rate, the combined event rate of cardiac death, MI and target lesion revascularization within 12 months. And incidence of composite events in cross over case of IVUS duing CTO intervention

SECONDARY OUTCOMES:
Incidence of MACE after stent implantation. | 24 months after CTO intervention
  1. Incidence of cardiac death, MI, TLR and ST for 9, 12 and 24 months after stent implantation.
  2. Binary restenosis, late loss, restenosis %, restenosis type and follow-up MLD on follow-up angiography 1 year after CTO intervention
  3. Subgroup analysis; : Among the IVUS guided intervention group, Non-IVUS giuded intervention group and total patient group,
     * To analyse difference of clinical outcome and angiographical outcome between Endeavor Resolute and Nobori stent.
     * To analyse change of Stenting distal part using IVUS parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Yang-Soo Jang, MD.PhD., Principal Investigator — Severance Hospital
Locations (1):
- Jang, Yang-Soo, Seoul, Seodaemun-gu/Sinchon-dong, South Korea

REFERENCES:
- [Derived] Kim BK, Shin DH, Hong MK, Park HS, Rha SW, Mintz GS, Kim JS, Kim JS, Lee SJ, Kim HY, Hong BK, Kang WC, Choi JH, Jang Y; CTO-IVUS Study Investigators. Clinical Impact of Intravascular Ultrasound-Guided Chronic Total Occlusion Intervention With Zotarolimus-Eluting Versus Biolimus-Eluting Stent Implantation: Randomized Study. Circ Cardiovasc Interv. 2015 Jul;8(7):e002592. doi: 10.1161/CIRCINTERVENTIONS.115.002592. PMID 26156151